CLINICAL TRIAL: NCT04660162
Title: Comparison of Laser Speckle Contrast Imaging and Laser Doppler Imaging
Acronym: LACOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maasstad Hospital (Other)
Responsible Party: Principal Investigator, Goksel Guven, Principle investigator, Research assistant in the Burn Unit of Maasstad Hospital, Maasstad Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: NL65747.101.18
Record Dates: First submitted 2020-11-22; First posted 2020-12-09 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Microcirculation
Keywords: microcirculation; laser speckle contrast imaging; laser doppler perfusion imaging; iontophoresis; comparison; flux
MeSH Terms: interventions — Iontophoresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm-1: Laser speckle contrast imaging (Experimental): (Perimed AB, Järfälla, Sweden)
  Interventions: Device: Iontophoresis; Other: Stepwise occlusion
- Arm-2: Laser Doppler perfusion imaging (Experimental): (Moor Instruments, Devon, UK)
  Interventions: Device: Iontophoresis; Other: Stepwise occlusion

INTERVENTIONS:
Device: Iontophoresis — By using the PeriIont (Perimed, Jarfalla, Sweden) device, 0.5 mL of a 10 mg/ml Sodium nitroprusside solution was used transdermally and ionised with a current strength of 200 µA for 1 minute.
Other: Stepwise occlusion — The upper arm was occluded for 30 seconds with a pneumatic cuff up to 50 mmHg, 80 mmHg, 110 mmHg, 140 mmHg, and 170 mmHg. The volunteer had rest for 5 minutes between each occlusion procedure.

SUMMARY:
The microcirculation plays a fundamental role in metabolic reactions and has been shown as an essential determinant in many clinical scenarios such as shock states, chronic and cardio-metabolic diseases. Microcirculation can be assessed directly using laser-based techniques and intravital microscopes. When combined with provocation tests, microvascular monitorization can be used to assess microvascular function.

Laser-based techniques are consist of two different methods named laser doppler imaging (LDI), laser speckle contrast imaging (LSCI). LSCI is a technique based on speckle contrast analysis that provides an index of blood flux. No need for skin contact, continuous and real-time assessment of the microcirculation led the LSCI to be broadly used in clinical practice. LDI is also a non-invasive diagnostic method used to measure the blood flux of tissue. The technique is based on measuring the doppler shift induced by moving red blood cells to the illuminating coherent light. Iontophoresis is one of the most commonly used provocation tests to study the endothelium in terms of endothelium-dependent and endothelium-independent vasodilation. Simultaneously with LDI and LSCI are used to follow and assess the skin blood flux during iontophoresis. Therefore, it provides a state to make a comparison between two different laser-based techniques in terms of flux characteristics.

The accurate assessment of burn depth is a critical step in the management of the burn-injured patient. Currently, LDI is the most widely used non-invasive measurement tool for assessing burn wounds and the only technique approved by the U.S. Food and Drug Administration. However, the LDI device is rather costly, cumbersome, and has a poor spatial resolution. LSCI measures perfusion in a similar way, but it provides high-quality images with a much higher spatial resolution. In addition, LSCI is much quicker, maneuverable, and able to assess larger skin areas. In order to use the LSCI technique in the clinical practice of burn-injured patients, as a first step, the linearity of LDI and LSCI should be shown. In this study, we aimed to compare LSCI and LDI with iontophoresis and stepwise occlusion technique. So, we will test the linearity of devices over a large range of blood flux values.

DETAILED DESCRIPTION:
Measurements of microcirculation were initiated upon the ethical consent was approved. 15 healthy volunteer were included in the study. All volunteers were asked for the existence of any symptoms for the on-going disease like flu, infectious disease, and chronic disease (Diabetes, hypertension, rheumatologic disorders, epileptic disorders, etc.). Once the volunteer met inclusion criteria, he/she became eligible for study. Volunteers were advised to beware from food and drink for at least two hours before measurement. Also, they were advised to come at least two hours after big meals like lunch or dinner. All the volunteers were evaluated at the same position (sitting and hand at heart level), room and temperature to provide equal standards. The volunteer had rest for at least 30 minutes in a semi-recumbent and extending leg position. The room temperature was 24-26C and checked with a thermometer intermittently. The door was closed to prevent air movement. Lights were switched off, and the curtains were closed to prevent the effect of light on devices. Once all the environmental conditions met, two investigators evaluated the volunteer. One investigator checked the volunteer's blood pressure, temperature, and heart rate.

A vacuum pillow was used to hold the arm stable during the procedure. Two different devices (laser speckle contrast imaging (LSCI) and laser doppler imaging (LDI)) were ready next to the volunteer. An appropriate intact skin area, inner side of the forearm were used for the investigation and both electrodes were attached. The skin surface was cleaned with alcohol or deionized water to remove remnants of cosmetics and creams with low conductivity. This helped to prevent spots with high current density that may result in local burns and non-specific vascular reactions. After peeling off the protective tape layer on the bottom of the Drug Delivery Electrode, the electrode was firmly attached to the skin. The Dispersive Electrode was placed approximately 10-15 cm from the Drug Delivery Electrode. Power supply was connected by attaching the electrodes to the leads. After lifting the lid of the Drug Delivery Electrode using the pointed tab, tip of the syringe was slided under the lid of the Drug Delivery Electrode and the Drug Delivery Chamber was filled with approximately 0.5 mL of a 10 mg/ml SNP solution. The drug was then delivered using cathodal iontophoresis for 1 minute with a current strength of 200 µA. The LDI and LSCI instruments are positioned so they can alternately measure the delivery site. Basal perfusion was measured with both instruments before starting iontophoresis. Subsequently, iontophoresis was started and measurements are made alternating between the two instruments. Therefore, we would be able to compare both devices in terms of supra-baseline flux values. When all measurements were finished, the electrodes removed from the patient and the Drug Delivery Electrode and the Dispersive Electrode was removed.

The second part of the study was performed as step-wise occlusion. The arm which was not used for iontophoresis test was used for step-wise occlusion. The baseline blood flux was followed for 2 minutes by LDI and LSCI. After 2 minutes, the upper arm was occluded for 30 seconds with a pneumatic cuff up to 50 mmHg, 80 mmHg, 110 mmHg, 140 mmHg, and 170 mmHg. Between each part, the volunteer had rest for 5 minutes to let the blood flux to turn the baseline. Once reaching to the planned pressure, LSCI and LDI devices were alternately be used to record blood flux. Therefore, we were able to compare both devices in terms of sub-baseline flux values.

All data were recorded in 2 external electronic storage, and the names of the volunteers were coded with numbers. Only main investigator was aware of who corresponds to which number. Results of Perimed and Moore Devices were analyzed with the software PIMsoft 1.5 (Perimed AB, Järfälla, Sweden), MoorLDI2-BI Burn's Software Version 4.0, respectively. Two investigators performed the analysis. If one investigator made the analysis, the other checked the results, as well.

ELIGIBILITY:
Inclusion Criteria:

* Should not have any disease at the time of procedure (including flu)
* Should not have any chronic disease
* Should not be under any medication
* Should not be smoker or ex-smoker
* Should not drink coffee or eat meal in two hours before the procedure
* Should not have an allergy to sodium-nitroprusside

Exclusion Criteria:

* Volunteer who does not meet any of the criteria above
* <18 years old
* Pregnant
* Refusal to participate in the study or demand to end study for any reason
* Hypersensitivity to sodium nitroprusside
* Broken or damaged skin surfaces
* Electrically-sensitive implanted devices such as cardiac pacemakers
* Maastad Ziekenhuis employers or collegues

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2018-12-17 (Actual)

PRIMARY OUTCOMES:
Comparison of Laser Speckle Contrast Imaging and Laser Doppler Imaging | 60 minutes
  Blood flux values of Laser Speckle Contrast Imaging device (Perimed AB, Järfälla, Sweden) and Laser Doppler Imaging device (Moor Instruments, Devon, UK) will be measured in a wide range of blood flux values and an equation formula will be described

SECONDARY OUTCOMES:
Creating common unit for Laser Speckle Contrast Imaging and Laser Doppler Imaging | 60 minutes
  Blood flux units will be measured and A new common and universal unit for laser based tecniques will be reported
Creating common color map for Laser Speckle Contrast Imaging and Laser Doppler Imaging | 60 minutes
  A new universal color code that is used by both Laser Doppler perfusion imaging and Laser speckle contrast imaging will be created based on the equation formula

CONTACTS AND LOCATIONS:
Overall Officials: Kees vd Vlies, MD, Study Director — Maasstad Hospital, Department of Burn Care; Can Ince, Phd, Study Director — Erasmus Medical Center, Department of Intensive Care
Locations (1):
- Maasstad Ziekenhuis, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sakr Y. Techniques to assess tissue oxygenation in the clinical setting. Transfus Apher Sci. 2010 Aug;43(1):79-94. doi: 10.1016/j.transci.2010.05.012. Epub 2010 Jun 17. PMID 20692624
- [Background] Briers JD. Laser Doppler, speckle and related techniques for blood perfusion mapping and imaging. Physiol Meas. 2001 Nov;22(4):R35-66. doi: 10.1088/0967-3334/22/4/201. PMID 11761081
- [Background] Tew GA, Klonizakis M, Crank H, Briers JD, Hodges GJ. Comparison of laser speckle contrast imaging with laser Doppler for assessing microvascular function. Microvasc Res. 2011 Nov;82(3):326-32. doi: 10.1016/j.mvr.2011.07.007. Epub 2011 Jul 22. PMID 21803051
- [Background] Stewart CJ, Frank R, Forrester KR, Tulip J, Lindsay R, Bray RC. A comparison of two laser-based methods for determination of burn scar perfusion: laser Doppler versus laser speckle imaging. Burns. 2005 Sep;31(6):744-52. doi: 10.1016/j.burns.2005.04.004. PMID 16129229
- [Background] Millet C, Roustit M, Blaise S, Cracowski JL. Comparison between laser speckle contrast imaging and laser Doppler imaging to assess skin blood flow in humans. Microvasc Res. 2011 Sep;82(2):147-51. doi: 10.1016/j.mvr.2011.06.006. Epub 2011 Jul 1. PMID 21745482
- [Background] Cordovil I, Huguenin G, Rosa G, Bello A, Kohler O, de Moraes R, Tibirica E. Evaluation of systemic microvascular endothelial function using laser speckle contrast imaging. Microvasc Res. 2012 May;83(3):376-9. doi: 10.1016/j.mvr.2012.01.004. Epub 2012 Jan 31. PMID 22326551
- [Background] Tesselaar E, Sjoberg F. Transdermal iontophoresis as an in-vivo technique for studying microvascular physiology. Microvasc Res. 2011 Jan;81(1):88-96. doi: 10.1016/j.mvr.2010.11.002. Epub 2010 Nov 9. PMID 21070791
- [Background] Wearn C, Lee KC, Hardwicke J, Allouni A, Bamford A, Nightingale P, Moiemen N. Prospective comparative evaluation study of Laser Doppler Imaging and thermal imaging in the assessment of burn depth. Burns. 2018 Feb;44(1):124-133. doi: 10.1016/j.burns.2017.08.004. Epub 2017 Oct 9. PMID 29032974
- [Background] Iredahl F, Lofberg A, Sjoberg F, Farnebo S, Tesselaar E. Non-Invasive Measurement of Skin Microvascular Response during Pharmacological and Physiological Provocations. PLoS One. 2015 Aug 13;10(8):e0133760. doi: 10.1371/journal.pone.0133760. eCollection 2015. PMID 26270037
- [Result] Ince C. The microcirculation is the motor of sepsis. Crit Care. 2005;9 Suppl 4(Suppl 4):S13-9. doi: 10.1186/cc3753. Epub 2005 Aug 25. PMID 16168069
- [Result] Klijn E, Den Uil CA, Bakker J, Ince C. The heterogeneity of the microcirculation in critical illness. Clin Chest Med. 2008 Dec;29(4):643-54, viii. doi: 10.1016/j.ccm.2008.06.008. PMID 18954699